CLINICAL TRIAL: NCT01030692
Title: Rivastigmine and Huperzine A as Treatments for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-24716; 1R01DA023624 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Cocaine Dependence; Cocaine Addiction; Cocaine Abuse; Substance Abuse
Keywords: Cocaine; Rivastigmine; Huperzine A
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Sugars; Rivastigmine; huperzine A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo capsules as control
  Interventions: Drug: Placebo
- Rivastigmine 3 mg (Active Comparator): Rivastigmine 3 mg
  Interventions: Drug: Rivastigmine 3 mg
- Rivastigmine 6 mg (Active Comparator): Rivastigmine 6 mg
  Interventions: Drug: Rivastigmine 6 mg
- Huperzine A 0.4 mg (Active Comparator): Huperzine A 0.4 mg
  Interventions: Drug: Huperzine A 0.4 mg
- Huperzine A 0.8 mg (Active Comparator): Huperzine A 0.8 mg
  Interventions: Drug: Huperzine A 0.8 mg

INTERVENTIONS:
Drug: Placebo — The placebo groups will receive the same dosage throughout the study.
  Other Names: Sugar pill
  Arms: Placebo
Drug: Rivastigmine 3 mg — The 3 mg rivastigmine group will receive 3 mg rivastigmine only in the evening of Day 1, 3 mg in the morning and 0 mg in the evening of Days 2-9, and 3 mg in the morning of Day 10.
  Other Names: Exelon
  Arms: Rivastigmine 3 mg
Drug: Huperzine A 0.4 mg — The 0.4 mg HupA group will receive 0.2 mg HupA only in the evening of Day 1, 0.2 mg in the morning and evening of Days 2-9, and 0.2 mg in the morning of day 10.
  Other Names: Huperzine
  Arms: Huperzine A 0.4 mg
Drug: Rivastigmine 6 mg — The 6 mg rivastigmine group will receive 3 mg rivastigmine only in the evening of Day 1, 3 mg in the morning and 0 mg in the evening of Days 2-5, 3 mg in the morning and evening of Days 6-9, and 3 mg in the morning of Day 10.
  Other Names: Exelon
  Arms: Rivastigmine 6 mg
Drug: Huperzine A 0.8 mg — The 0.8 mg HupA group will receive 0.2 mg HupA only in the evening of Day 1, 0.2 mg in the morning and evening of Days 2-5, 0.4 mg in the morning and evening of Days 6-9, and 0.4 mg in the morning of Day 10.
  Other Names: Huperzine
  Arms: Huperzine A 0.8 mg

SUMMARY:
The purpose of this study is to determine the safety and effects of rivastigmine and huperzine A (HupA), potential treatments for cocaine abuse, when used before experimental administration of cocaine, on a number of physical and psychological measures.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the interactions between cocaine and oral rivastigmine and between cocaine and oral huperzine A (HupA).

The following Specific Aims are proposed: 1. Among cocaine-dependent, non-treatment seeking participants, to establish the ability of rivastigmine (3 or 6 mg, daily) or HupA (0.4 or 0.8 mg, daily), as compared to placebo, to reduce cocaine-induced craving (0, 20, and 40 mg, IV) and to reduce reinforcing effects produced by cocaine (20 mg, IV/infusion). Hypothesis. Relative to placebo-treated participants, treatment with rivastigmine or HupA will reduce cocaine-induced craving and choices for cocaine.

2. To determine the safety of rivastigmine and HupA in cocaine-dependent participants who receive cocaine in a laboratory setting. Hypothesis 2A. Relative to placebo-treated participants, treatment with rivastigmine or HupA will not increase the adverse events produced by cocaine. Hypothesis 2B. Relative to placebo-treated participants, treatment with rivastigmine or HupA will reduce cocaine-induced increases in heart rate and blood pressure.

3. To determine the effects of AChE inhibition on plasma levels of cocaine and cocaine metabolites. Hypothesis 3A. Relative to placebo-treated participants, treatment with rivastigmine, but not HupA, will be associated with increased plasma levels of cocaine. Hypothesis 3B. Relative to placebo-treated participants, treatment with rivastigmine, but not HupA, will be associated with increased formation of ecgonine and benzoylecgonine, and decreased formation of ecgonine methylester.

4. a) provide a more frequent measure of heart rate (15 sec vs. 5 minutes) and b) measure a new dependent variable, physical activity, on days with and without cocaine exposure.

Public Health Significance: Cocaine abuse is an important health problem that is associated with serious medical, psychiatric, social, and economic consequences. No medications are currently available for prevention of relapse in patients who are addicted to cocaine, and compounds such as rivastigmine and HupA are predicted to be useful for this indication. The testing of HupA is particularly exciting since it has antioxidant and neuroprotective properties that may also contribute to its efficacy as a treatment medication for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Be a cocaine-dependent volunteer who is non-treatment-seeking
* Meets DSM-IV criteria for cocaine dependence as determined by SCID, and has provided at least one cocaine-positive urine specimen within the 2 weeks prior to enrollment
* Be male or female, between 18 and 55 years old
* Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures
* Female subjects must be non-nursing and postmenopausal, have had a hysterectomy, undergone tubal ligation, or have a negative pregnancy test and agree to use one of the birth control methods below
* Agreeable to conditions of the study and likely to complete schedule of interventions and measures
* Has medical history, physical exam, and screening laboratory results that demonstrate no contraindication to participation

Exclusion Criteria:

* Has a history of a medical adverse reaction to cocaine or other psychostimulants, including loss of consciousness, chest pain, cardiac ischemia, or seizure
* Has a current psychiatric disorder other than cocaine abuse or dependence, including major depression, bipolar disorder, schizoaffective disorder, schizophrenia, organic brain disease, or dementia
* Meets DSM-IV criteria for dependence to opiates, benzodiazepines, alcohol, or other sedative-hypnotics
* Receiving opiate-substitution therapy (methadone, LAAM, or buprenorphine) within 2 mo's of enrollment
* Has a current or past history of seizure disorder, including alcohol- or psychostimulant- related seizures, febrile seizures, or family history of seizure disorder
* Has a diagnosis of adult (i.e., 21 years or older) asthma, or chronic obstructive pulmonary disease, including a history of acute asthma within the past two years, and those with current or recent (with the past two years) treatment with an inhaled or oral b-adrenergic agonist
* Has had head trauma that resulted in neurological sequelae (e.g., loss of memory for greater than 5 min or that required hospitalization)
* Has an unstable medical condition, which, in the judgment of investigators, would make participation hazardous, including, but not limited to, AIDS, acute hepatitis, active TB, unstable cardiac disease, unstable diabetes, hepatic or renal insufficiency (serum bilirubin or creatinine exceeding 1.5 the upper limit of normal, respectively)
* Be pregnant or lactating (nursing), or a fertile woman not practicing adequate methods of contraception or planning to become pregnant within one month of conclusion of the study
* Has current suicidal ideation or plan as assessed by SCID or MINI interview
* Has clinically significant ECG abnormalities, including QTc interval prolongation >450 ms in men or >480 ms in women
* In the opinion of the PI, be expected to fail to complete the study protocol due to probable incarceration or relocation from the clinic area
* Has clinically significant laboratory values (outside of normal limits), in the judgment of the PI
* Is on parole, probation or has any legal obligations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The effects of rivastigmine or huperzine A and cocaine on cardiovascular measures | 10 days
  Before and after each cocaine infusion, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on rivastigmine or HupA relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, changes in cocaine PKs, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of rivastigmine or huperzine A and cocaine on subjective measures | 10 days
  The ability of rivastigmine (3 or 6 mg, daily) or HupA (0.4 or 0.8 mg, daily), as compared to placebo, to reduce cocaine-induced craving (0, 20, and 40 mg, IV) and to reduce reinforcing effects produced by cocaine (20 mg, IV/infusion) will be measured by: 1. VAS, Adjective Scales, and MCQ; 2. Choices for cocaine vs. money in the self-administration assay.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, II, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States